CLINICAL TRIAL: NCT04515160
Title: Correlation of Clinical Frailty Scale and Modified Frailty Index in Intensive Care Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Bahar SAKIZCI UYAR, medical doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: 92/04
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Clinical Frailty Scale — Clinical fragility scale will be recorded in the first 24 hours of intensive care admissions.
Diagnostic Test: Modified Frailty Index — Modified Frailty Index will be recorded in the first 24 hours of intensive care admissions.

SUMMARY:
The purpose of our study is to evaluate the correlation of the Clinical Frailty Scale, which is a judgment-based measure, and the Modified Frailty Index, which interrogates the patient's current diseases, in the frailty assessment of intensive care patients and the effect on the estimation of mortality, mechanical ventilation need, intensive care stay, hospital stay and discharge status.

ELIGIBILITY:
Inclusion Criteria:

* intensive care patients

Exclusion Criteria:

* patients with a life expectancy of less than 24 hours
* Do not speak Turkish

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: intensive care patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Frailty | in the first 24 hours of intensive care admissions
  the correlation of the Clinical Frailty Scale, which is a judgment-based measure, and the Modified Frailty Index, which interrogates the patient's current diseases, in the frailty assessment of intensive care patients

SECONDARY OUTCOMES:
mortality | the patient will be monitored for 1 year and the exitus time will be recorded
  effect of the clinical frailty scale and modified farilty index on the estimation of mortality
intensive care stay | the patient will be monitored for 1 year and the intensive care stay will be recorded
  effect of the clinical frailty scale and modified farilty index on the estimation of intensive care stay
discharge status | the patient will be monitored for 1 year and the discharge status will be recorded
  effect of the clinical frailty scale and modified farilty index on the estimation of discharge status

CONTACTS AND LOCATIONS:
Locations (1):
- DiskapiYBERH, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No